CLINICAL TRIAL: NCT02731118
Title: Antisecretory Factor (AF) Effects on Intraocular-pressure: a Placebo-controlled Randomised Study
Brief Title: Antisecretory Factor (AF) Effects on Intraocular-pressure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty recruiting patients and no effect on preliminary analysis
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Enping Chen, MD PhD, St. Erik Eye Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sal/2016
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma
Keywords: glaucoma; intraocular pressure lowering treatment; antisectory factor (AF); Salovum
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo and Salovum (Experimental): 6 times 4 gr placebo/Salovum day 1-2, 5 times 4 gr placebo/Salovum day 3-5, 4 times 4 gr placebo/Salovum day 6-14
  Interventions: Dietary Supplement: Salovum; Dietary Supplement: Placebo
- Salovum and placebo (Experimental): 6 times 4 gr Salovum/placebo day 1-2, 5 times 4 gr Salovum/placebo day 3-5, 4 times 4 gr Salovum/placebo day 6-14
  Interventions: Dietary Supplement: Salovum; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Salovum — AF-enriched egg yolk
Dietary Supplement: Placebo — egg yolk

SUMMARY:
Glaucoma is a complex and chronic eye disease which damages the optic nerve. One of the main risk factors for the progression of glaucoma is IOP.

The aim of the study is to examine if Salovum, an anti-secretory factor (AF), can reduce the level of the intraocular pressure (IOP) in the eye of patients affected by glaucoma.

Anti-secretory factor (AF) is an endogenous protein which controls the transport of water and ions across the cell membrane. AF plays an important part in the immune system and has an anti-secretory and anti-inflammatory effect.

The investigators' hypothesis is that Salovum can restore a normal salt-water balance in the eye, which in turn would lower the IOP. This would eliminate or reduce the risk of subsequent visual impairments/neurological damage.

DETAILED DESCRIPTION:
The aim of the study is to examine if Salovum, an anti-secretory factor (AF), can reduce the level of the intraocular pressure (IOP) in the eye of patients affected by glaucoma.

Glaucoma is a complex and chronic eye disease which damages the optic nerve. Beginning at the periphery of the vision field, it often progresses very slowly, which means that the patients consult a doctor only when damages have become very large. Glaucoma requires a lifelong medical treatment. Regardless of the medical treatment, damaged nerve fibers will never regenerate. An early onset of the medical treatment is crucial to avoid the progression of the disease which, if not treated, would also affect the central vision, resulting in patients with severe handicap.

One of the main risk factors for glaucoma is elevated IOP and treatment is aimed to reduce its progression by IOP lowering. About 10-15 % of glaucoma patients following a medically correct treatment respond poorly or not at all to the medicines, leading to a progressive loss of the visual field and an increasingly defective eyesight.

Anti-secretory factor (AF) is an endogenous protein which has been characterized in vivo and in vitro. AF is a part of the proteasome and controls the transport of water and ions across the cell membrane. AF plays an important part in the immune system and has an anti-secretory and anti - inflammatory effect in vivo along with complementary substances, primarily c3C. Researchers have chemically characterized and cloned AF's cDNA and shown that the active part (anti-secretory and anti-inflammatory) is located in the amino terminal portion of the protein. The exact mechanisms behind AF's regulatory effect on the secretory / inflammatory progress, however, is largely unknown, but AF is probably involved in the liquid transport mechanisms in the cell pathway.

AF has been detected in most of the body tissues, plasma, breast milk, bile and faeces. In healthy individual, AF occurs principally in an inactive form, but AF can be activated by a disease, e.g. the toxin-induced diarrhea. The transition from inactive to active AF contributes to the normalization of the intestinal secretion and diarrhea decreases or ceases. In human beings, AF therapy has reduced disease symptoms such as ulcerative colitis, Crohn's disease, Meniere's disease, mastitis (inflammation of the mammary gland ) and during diarrhea conditions of different genesis. AF treatment has been particularly successful in the treatment of children's diarrhea and is routinely used in Pakistan. No side effects of therapy have so far been reported. Experiences in rats have also shown that AF is effective in lowering the pressure in the tissue tumors (breast cancer), lowering the elevated intracranial pressure that arises in connection with virus-induced inflammation of the brain (herpesvirus type 1), reducing the pressure caused by mechanical brain damage that mimic stroke (frost damage).

By giving egg-producing hens special feed, hens' own production of AF is stimulated. The high content of AF is specifically reflected in the egg yolk with a level about 10,000 times higher than in normal eggs. The AF enriched egg yolk is subjected to spray-drying and sealed in bags containing 4 gr each. This product is named Salovum and has been registered as a food for specific medical purposes through the regulatory authorities in the EU. However, Salovum cannot be used in patients with diagnosed or suspected with egg allergy.

The investigators' hypothesis is that Salovum can restore a normal salt-water balance in the eye, which in turn would lower the IOP. This would eliminate or reduce the risk of subsequent visual impairments/neurological damage. It is in this context important to point out that the intake of Salovum counts as food and does not in any way interfere with the conventional medical management of glaucoma.

Fifty glaucoma patients who despite adequate medication need additional IOP lowering will be recruited. Participants will be randomly divided into 2 groups with 25 patients each and will be treated according to the following:

* one group begins with Salovum during 2 weeks and then take a placebo for another 2 weeks
* one group begins with placebo for 2 weeks and then takes Salovum 2 weeks.

Dosage: Salovum is dissolved in juice or water and may give rise to a certain satiety. Each bag contains 4 gr of dried egg yolk. The first 2 days, the patients will take one bag of Salovum or placebo 6 times a day , then a bag 5 times daily for 3 days and finally a bag 4 times daily for 9 days.

The eye which has the highest IOP will be selected. If both eyes have the same IOP, the right eye will be chosen. IOP will be measured according to Goldmann applanation tonometry five times during the study period. IOP will be measured three times per session and all three measurements will be used for statistical analysis. IOP will also be measured with a self-tonometer by the patients themselves 5 times daily.

Patients will get more detailed information about handling the self-tonometer from study staff. All results will be stored at St Erik Eye Hospital in a computer system with limited access.

During the study, patients will continue to take their glaucoma treatment as usual. Except for drinking Salovum and measuring their IOP, no new routine will encounter.

As the study will compare placebo (egg yolk with a low level of AF) with active treatment (Salovum with a high dose of AF) within a sick patient population, no healthy subjects will be included in the study.

If an IOP lowering effect is achieved with Salovum, the investigators will discuss with the patient how treatment should be continued. If no effect is obtained, patients will continue with their usual medical treatment only.

ELIGIBILITY:
Inclusion Criteria:

* open angle glaucoma, ocular hypertension

Exclusion Criteria:

* other types of glaucoma, other types of ocular comorbidity, previous intra-ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 2 weeks
  IOP lowering effect of treatment or placebo over 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Enping Chen, MD PhD, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St Erik Eye Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No